CLINICAL TRIAL: NCT00495352
Title: 1. The Pharmacogenetic Study of Interaction Among Antipsychotics, Readiness to Change, and Pharmacological Intervention for Smoking Cessation Among Schizophrenic Patients 2. Stages of Change and Outcomes of Nicotine Replacement Therapy in Chronic Schizophrenic Patients
Brief Title: The Pharmacogenetic Study , Readiness to Change, and Pharmacological Intervention for Smoking Cessation in Schizophrenia
Acronym: PSIAARP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yu-Li Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Yu-Li Hospital, Yu-Li Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-095-PP-05A
Record Dates: First submitted 2007-06-30; First posted 2007-07-03 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Tobacco Dependence; Schizophrenia
Keywords: Schizophrenia; NRT; Bupropion; Stages of change
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia | interventions — Nicotine Replacement Therapy; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-dose NRT, Low-dose NRT, bupropion (Active Comparator)
  Interventions: Drug: Hihg-doseNRT, Low-dose NRT, bupropion

INTERVENTIONS:
Drug: Hihg-doseNRT, Low-dose NRT, bupropion

SUMMARY:
Cigarette smoking represents a major health problem for patients suffering from schizophrenia. Compared to the general population, schizophrenic patients are significantly more likely to be addicted to nicotine. They also are more likely to be heavy smokers, and tend to be exposed disproportionately to nicotine and other harmful ingredients in the cigarette because of the observed tendency to smoke down to the very end. Further, smoking in these patients may be associated with a higher risk for developing tardive dyskinesia All of these factors render schizophrenic patients a particularly vulnerable group for the detrimental effects of tobacco-related medical problems. Currently, there is little information available regarding the efficacy and utility of smoking cessation treatment methods, as well as factors that may predict patients' response to such treatments.

An important related issue is the influence of smoking, and its cessation, on the effects of the medications most of these patients rely upon for the control of their psychiatric symptoms. Although smoking has long been known to significantly alter the metabolism, and thus the effects, of most antipsychotics, the extent and clinical significance of these influences have rarely been assessed. It is unclear to what extent smoke cessation (as well as initiation) changes the side effect profiles of these medications, and whether such changes contribute towards the difficulties in patients' ability and/or willingness to stop smoking.

In addition, except pharmacological intervention, readiness to change may be an important factor affecting the outcomes of smoking reduction. Prochaska et al proposed the concept of stages of change to predict the response of quitting behavior for substance use. A lot of evidence support the stronger of readiness of change, the higher successful rate of quitting can be reached. Yet these results are largely found in many non-pharmacological intervention and smoking cessation programs for general population. Till now, no available study solely focus readiness of change quitting smoking behavior in NRT treatment for chronic schizophrenic patients. Thus, we have an a great interest in examining the association between the stages of change and the outcomes of smoking-cessation along with reduction among schizophrenic patients receiving transdermal nicotine patches.

In order to begin addressing these important issues, this application proposes to utilize state-of-the-art methodologies derived from the field of pharmacogenetics, molecular biology and clinical trials, to (1) examine short-term and long-term efficacy of standard treatment methods, such as the use of nicotine patches, in this population; (2) identify factors that might predict treatment responses; and, (3) examine the interactions between smoking and the effect of antipsychotics, as well as how such interactions might affect smoking cessation. (4) to examine the predictive value of the stages of change on smoking cessation and reduction outcomes in schizophrenic patients receiving different doses of nicotine replacement therapy (NRT) and bupropion as implemented in a randomized trial.

DETAILED DESCRIPTION:
Specific Aims

Accordingly, this proposal aims at testing the following major hypotheses:

1. Nicotine patch therapy and bupropion are effective in smoke cessation among motivated psychiatric outpatients with schizophrenia.

1a. High dose nicotine patch therapy is significantly more effective in inducing smoke cessation than regular dose nicotine patch therapy.

1b. Nicotine patch therapy and bupropion are more effective in inducing smoke cessation in those treated with "atypical" neuroleptics as compared to those treated with "typical" neuroleptics.

2. Response to nicotine patch therapy is associated with genetic polymorphisms of DRD2, dopamine transporter (DAT; SLC6A3), CYP2A6 and CYP2D6 genes.

3. Smoke cessation is associated with a significant decrease in the activity of CYP1A2, as well as a significant increase in the steady-state concentration of the neuroleptics received by the patients. This will lead to an increased incidence of treatment emergent side effects, which may be controlled by neuroleptic dose adjustment.

4. patients in the stage of preparation or contemplation (stronger readiness to quit smoking) are more likely to reduce smoking and stop smoking than those in the stage of precontemplation (weaker readiness to quitting smoking).

ELIGIBILITY:
Inclusion Criteria:

* Competent volunteers completing consent form
* Schizophreniform, schizoaffective,or psychotic disorder NOS based on DSMIV

Exclusion Criteria:

* Severe life-threatening physical condition
* Pregnancy
* Fluroxamine treatment in the past 2 weeks
* Allergy to nicotine or caffeine

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-01; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence of abstinence | 8 weeks after the initiation of this trial

SECONDARY OUTCOMES:
smoking reduction more than 50% and 25% | 8 weeks after the initiation of this trial

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD, Ph.D, Study Director — General Clinical Research Center, YuLi hospital
Locations (1):
- Yuli hospital, DOH, Yuli Townhsip, Taiwan